CLINICAL TRIAL: NCT06822231
Title: Clinical Protocol for a Pragmatic Trial on a High-Tech Rehabilitation Pathway for Acute Adult Neuromuscular Diseases (Fit4MedRob-Acute MND Project)
Brief Title: High-Tech Rehabilitation Pathway for Acute Adult Neuromuscular Diseases - Fit4MedRob-Acute MND Project
Acronym: Fit4MR-AcMND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Modena (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024_0053110; PNC0000007 (Other Grant/Funding Number: Ministry of University and Research)
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness Myopathy; Guillain Barré Syndrome; Critical Illness Polyneuromyopathy (CIPNM)
Keywords: high-tech rehabilitation; acute neuromuscular diseases; robotic platform
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic treatment group (Active Comparator): In this arm, patients will be divided into 3 treatment types based on their Berg Balance Scale (BBS) score at the time of randomization. Phase 1 (BBS <= 20) involves treatment with a robotic verticalization system (ERIGO) and action observation training with a virtual reality device.
  Phase 2 (21 < BBS < 40) involves treatment with a robotic verticalization system (ERIGO), action observation training with a virtual reality device, and proprioceptive exercises on robotic platforms (e.g. GEA MASTER or PROKIN Technobody).
  Phase 3 (BBS >= 41) involves motor and cognitive exercises using virtual reality device, proprioceptive exercises on robotic platforms (e.g. GEA MASTER or PROKIN Technobody), and aerobic exercises on a robotic treadmill (e.g. Walkerview Technobody).
  Interventions: Device: High-tech rehabilitative treatment
- Control group (Other): The patients will receive the traditional rehabilitative treatment according to the good clinical practice according to the Diagnostic, Therapeutic and Care Pathways of each center involved
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Device: High-tech rehabilitative treatment — Robotic Verticalization System (e.g., Erigo): Assists in regaining upright posture and mobility.
  Virtual Reality (e.g., VRRS Evo): Provides an engaging and immersive environment for cognitive and motor exercises.
  Stabilometric Platform (e.g., Gea Master or Prokin Technobody): Used for balance and postural control training.
  Treadmill System (e.g., Walkerview Technobody): Used for aerobic exercises with gait analysis and feedback
  Arms: Robotic treatment group
Other: Rehabilitation — Traditional rehabilitative treatment
  Arms: Control group

SUMMARY:
The goal of this study is determine if a high-tech rehabilitation circuit is more effective than usual rehabilitation methods in improving functional outcome, particularly balance control, for patients with acute neuromuscolar diseases. The main question it aims to answer is:

Are high-tech rehabilitation interventions, including robotic systems, virtual reality, and stabilometric platforms, more effective than traditional rehabilitation methods in improving balance, motor function, fatigue levels, sarcopenia, cognitive engagement, and overall quality of life in patients with acute neuromuscular diseases (NMDs)? Researchers will compare a robotic treatment group, that consists in an high-tech rehabilitation, with a control group, that will receive the traditional rehabilitative treatment.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy of a novel rehabilitation protocol integrating advanced technologies in the treatment of acute neuromuscular diseases (NMDs).

Background: NMDs affect muscle function and are directly controlled by the nervous system. Traditional rehabilitation often falls short in addressing the multifaceted needs of NMD patients. This gap underscores the necessity for innovative rehabilitation approaches that can significantly enhance the quality of life and optimize recovery outcomes following acute events.

Methods: The protocol integrates advanced technologies to address the rehabilitation needs of patients with acute NMDs. It utilizes robotic systems to ensure consistent and precise movement, virtual reality for immersive and engaging therapy, and stabilometric platforms to enhance balance training. The focus is on acute NMDs such as Guillain-Barré Syndrome (GBS), Critical illness myopathy (CIM) and polyneuropathy (CIP), either individually or in combination (CIP/CIM). The approach emphasizes rapid rehabilitation to maximize recovery outcomes.

Study Design: An interventional, randomized, superiority case-control study with a parallel assignment. The trial aims to compare the efficacy of high-tech rehabilitation methods against conventional treatments in improving patient outcomes.

Outcome Measures: To assess the improvement at least 10 points in balance measured using the Berg Balance Scale (BBS) from baseline to the end of the treatment period comparing the high-tech rehabilitation circuit with standard rehabilitation protocol.

Conclusion: This protocol seeks to determine if high-tech rehabilitation interventions can outperform traditional methods in acute NMDs. By doing so, it aims to potentially establish a new global standard for the care of patients with NMD care.

ELIGIBILITY:
Inclusion Criteria:

* Adults with ages ranging from 18 to 80 years.
* Patients with a confirmed diagnosis of acute/subacute neuromuscular diseases (e.g. GBS, CIM, CIP)
* Time of onset ranging from 15 to 30 days
* Patients with lower limb strength (Medical Research Council or MRC) >=2 in at least two of the flexor and extensor muscles of the following joints: hip, knee and ankle
* Possibility of obtaining informed consent

Exclusion Criteria:

* Patients with unstable medical conditions (e.g. severe cardiovascular diseases, such as "New York Heart Association" - NYHA=4, respiratory distress not compensated by ventilation) that could interfere, in the clinician's judgment, with their ability to safely participate in the study or to perform the assessments related to the protocol.
* Patients currently participating in other clinical trials that could interfere with this study.
* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Berg Balance Scale | At the end of treatment at day 60
  Improvement in balance measured by the Berg Balance Scale (BBS), with a target improvement of at least 10 points from baseline to the end of the treatment period. BBS is used to objectively determine a patient's ability (or inability) to safely balance during a series of 14 tasks; each task ranks from 0 to 4, with a total score of 56. Higher score indicates the higher level of function.

SECONDARY OUTCOMES:
Change from baseline in Modified Barthel Index | At day 15, at day 30, at day 45, at day 60
  Modified Barthel Index (MBI). The MBI is an adaptation of the original Barthel Index, designed to assess a patient's ability to perform activities of daily living (ADLs) and their level of independence. The MBI evaluates ten specific functions: Feeding, Bathing, Grooming, Dressing, Bowel control, Bladder control, Toileting, Transfers (e.g., bed to chair), Mobility (e.g., walking or wheelchair use), Stair climbing. Each item is scored on a 5-level ordinal scale. Interpretation: 0-20, Total dependency; 21-60, Severe dependency; 61-90, Moderate dependency; 91-99, Slight dependency; 100, Independence
Change from baseline in Trunk Control Test | At day 15, at day 30, at day 45, at day 60
  Trunk Control Test (TCT) for non-ambulatory patients. The TCT is a clinical assessment tool used to evaluate trunk movement control in patients, particularly those who have suffered a stroke or other neurological disorders. The TCT measures four specific movements: 1) Rolling to the weak side: The patient rolls from a supine position to their weaker side; 2) Rolling to the strong side: The patient rolls from a supine position to their stronger side; 3) Balance in a sitting position: The patient sits on the edge of a bed or table without support for at least 30 seconds; 4) Sitting up from lying down: The patient moves from a lying to a sitting position. Each movement is scored on a scale from 0 to 25, with a total possible score of 100. Higher scores indicate better trunk control (Collin & Wade 1990)
Change from baseline in 2-Minute Walk Test | At day 15, at day 30, at day 45, at day 60
  2-Minute Walk Test (2MWT) for ambulatory patients. The Two-Minute Walk Test (2MWT) is a simple and quick assessment used to measure a person's walking endurance and functional mobility. It is based on the measurement of the distance that a person can walk in two minutes. The individual is instructed to walk as far as possible in two minutes, typically along a marked course. Assistive devices can be used if needed, but should be kept consistent across tests. The total distance walked in meters or feet is recorded
Change from baseline in Modified Erasmus GBS Outcome Score | At the end of treatment at day 60
  Modified Erasmus GBS Outcome Score (mEGOS) for Guillain-Barrè Syndrome patients: is a clinical prediction model used to estimate the likelihood of a patient with GBS being unable to walk independently six months after disease onset. This score is calculated based on three key factors: 1) Age at onset of neurological symptoms; 2) Preceding diarrhea before the onset of symptoms; 3) Severity of muscle weakness, assessed using the Medical Research Council sum score. The mEGOS provides a score ranging from 0 to 12, with higher scores indicating a higher risk of walking inability
Change from baseline in Handgrip strenght test | At day 15, at day 30, at day 45, at day 60
  Maximal isometric handgrip strength for both right and left hands will be measured using a digital handgrip dynamometer in units of kg/f in the standardized position recommended by the American Society of Hand Therapists, that is, sitting in a chair with a 90° backrest and 90° elbow flexion of the hand to be evaluated. Each participant exerted three trials of 3 s of maximal isometric handgrip strength alternatively for the right and left hands, with a rest period of 180 s between trials and considering the best performance of the three trials for statistical analysis
Change from baseline in Isometric muscles strenght | At day 15, at day 30, at day 45, at day 60
  Isometric muscle strength, measured in kg, was assessed using a manual hand-held dynamometer (HHD) at the deltoid, biceps brachii, triceps brachii, wrist flexor, and wrist extensor for the upper limbs bilaterally; thigh flexor, knee extension, knee flexion, dorsiflexion, and plantarflexion for the lower limbs bilaterally
Change from baseline in Numeric Rating Scale | At day 30 and day 60
  Measured using the Numeric Rating Scale (NRS). The NRS for fatigue is a simple and widely used tool to assess the intensity of fatigue. It helps patients communicate their fatigue levels to healthcare providers effectively. The NRS typically uses an 11-point scale ranging from 0 (no fatigue) to 10 ("the worst fatigue imaginable"). Patients are asked to rate their fatigue by selecting a number that best represents their pain intensity at that moment.
Change from baseline in 12-Short Form-12 Survey | At day 30 and day 60
  It will be used the 12-Item Short Form Survey (SF-12). The SF-12 is a self-reported questionnaire designed to measure health-related quality of life. It is a shortened version of the SF-36, created to reduce the burden on respondents while still providing reliable and valid results. The SF-12 covers eight health domains: Physical functioning; Role-physical (limitations due to physical health problems); Bodily pain; General health; Vitality (energy and fatigue); Social functioning; Role-emotional (limitations due to emotional problems); Mental health (psychological distress and well-being). The survey produces two summary scores: Physical Component Summary (PCS) and Mental Component Summary (MCS). These scores are norm-based, with a mean of 50 and a standard deviation of 10. Scores above 50 indicate better-than-average health-related quality of life, while scores below 50 suggest below-average health
Change from baseline in Technology Assisted Rehabilitation Patient Perception Questionnaire | At day 30, at day 60
  To assess the patient perception of the technology assisted rehabilitation using the Technology Assisted Rehabilitation Patient Perception Questionnaire (TARPP-Q). The TARPP-Q consists of 10 questions with multiple choice answers, totalling 29 items. The Questionnaire assesses patients' personal experiences and perceptions of technology assisted rehabilitation, including aspects like usability, positive attitude, hindrance perception, and distress.

OTHER OUTCOMES:
Change from baseline in Insulin Growth Factor 1 and free Insulin Growth Factor 1 | At day 15, at day 30, at day 60
  Will be measured these biomarkers in order to assess the levels changes during the treatment. Serum level will be measured in nanogram/milliliter
Change from baseline in Neurofilament-Light chain | At day 15, at day 30, at day 60
  Will be measured this biomarker in order to assess the levels changes during the treatment. Plasma level will be measured in picogram/milliliter.

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Istituti Clinici Scientifici Maugeri, Bari
  - IRCCS Azienda Ospedaliera Universitaria San Martino - Genova, Genova
  - Istituti Clinici Scientifici Maugeri IRCCS, Milan Institute, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Istituti Clinici Scientifici Maugeri, Montescano
  - Istituti Clinici Scientifici Maugeri, Pavia
  - Fondazione Don Carlo Gnocchi Onlus, Roma
  - Istituti Clinici Scientifici Maugeri, Telese Terme

IPD SHARING:
Plan to Share IPD: No